CLINICAL TRIAL: NCT00037284
Title: Behavioral and Immunological Factors in Coronary Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1159; R01HL066149 (NIH)
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2008-07

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Depression
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Depression

SUMMARY:
To explore the immune/inflammatory processes as pathways between depression/exhaustion and coronary artery disease (CAD) progression.

DETAILED DESCRIPTION:
BACKGROUND:

Recent studies demonstrate that the immune system plays an important role in coronary artery disease (CAD). Research also shows that psychological factors such as major depression and acute mental stress are involved in the clinical progression of CAD. Depression is associated with higher levels of immune parameters that play a role in CAD (cytokines, markers of low grade inflammation, infectious pathogen burden, and adhesion molecules), and most of these measures also increase in response to acute physical and mental stress. The pathophysiological mechanisms linking depression and mental stress with adverse cardiovascular outcomes may therefore be mediated by immunological factors.

DESIGN NARRATIVE:

The study examines clinical outcomes in patients who undergo percutaneous coronary revascularization, because a major problem remains the frequent (20 percent-40 percent) occurrence of coronary restenosis and new cardiac events in the six months after the intervention. These adverse outcomes have substantial impact on the costs of medical care and patients' quality of life. Since previous research has not examined the role of behaviorally-induced changes in immune parameters in the prediction of CAD progression, the following immunological measures will be examined: cytokines (IL-1B, IL-4, IL-6, IFNy, TNFa), acute phase proteins (CRP, fibrinogen), lymphocyte counts and differential, adhesion molecules (ICAM-1, LFA, L-selectin), and a composite measure of pathogen burden (CMV, H. pylori, C. pneumoniae). Using a longitudinal design, this project will determine the time course of changes in depression and changes in immune parameters. Moreover, the present study will determine the contribution of behavioral and immunological factors in the clinical progression of coronary disease following coronary angioplasty. These data may therefore improve the identification of patients at risk for recurrent cardiac events and restenosis after coronary angioplasty, and provide further understanding of the pathophysiological mechanisms involved in coronary disease progression.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Willem Kop — Uniformed Services University of the Health Sciences

REFERENCES:
- [Background] Kop WJ, Gottdiener JS, Tangen CM, Fried LP, McBurnie MA, Walston J, Newman A, Hirsch C, Tracy RP. Inflammation and coagulation factors in persons > 65 years of age with symptoms of depression but without evidence of myocardial ischemia. Am J Cardiol. 2002 Feb 15;89(4):419-24. doi: 10.1016/s0002-9149(01)02264-0. PMID 11835923
- [Background] Kop WJ. The integration of cardiovascular behavioral medicine and psychoneuroimmunology: new developments based on converging research fields. Brain Behav Immun. 2003 Aug;17(4):233-7. doi: 10.1016/s0889-1591(03)00051-5. PMID 12831824
- [Background] Kop WJ, Gottdiener JS. The role of immune system parameters in the relationship between depression and coronary artery disease. Psychosom Med. 2005 May-Jun;67 Suppl 1:S37-41. doi: 10.1097/01.psy.0000162256.18710.4a. PMID 15953799